CLINICAL TRIAL: NCT04844827
Title: Creation of a Pleural Carcinomatosis Tissue Bank
Brief Title: Pleural Carcinomatosis Tissue Banking
Acronym: TICP
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0116; 2021-A00761-40 (Other: ID-RCB)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Pleural Effusion, Malignant
Keywords: Malignant pleural effusion; pleural carcinomatosis; pleural metastasis; tissue banking
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Between 3 and 5 pleural biopsies and 5 blood samples for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malignant pleural effusion: Patients with malignant pleural effusion who underwent pleural biopsies and blood tests under general anesthesia
  Interventions: Genetic: Conserving routinely performed pleural biopsies in our biological resources center to realize multiomics and bioinformatics analyzes secondarily

INTERVENTIONS:
Genetic: Conserving routinely performed pleural biopsies in our biological resources center to realize multiomics and bioinformatics analyzes secondarily — Interventions will consist of a diagnostic and symptomatic videothoracoscopy in patients with pleural metastasis under general anesthesia, as part of a standard of care procedure. Fragments of these pleural biopsies (one for routine diagnosis and two for scientific purposes) will enrich the biocollection. Five blood samples will be taken at the time of surgery (3 to 5 ml / tube). These biological samples will be stored in the HCL CRB tumor bank. At the same time, patient demographic data will be collected and anonymized. In the long term, the biological material will be used by IARC for carrying out multi-omics and bioinformatics analyzes

SUMMARY:
Malignant pleural effusion is a common evolution of various cancers and is associated with poor prognosis and quality of life. About 28% of patients with primary malignancy will develop pleural metastasis. Malignant pleural effusion mostly occurs in lung, breast, ovarian and gastric cancers. Median survival ranges from 3 to 13 months according to primary malignancy. Currently, the therapeutic approach is mainly palliative with videothoracoscopic talc pleurodesis or indwelling pleural catheters insertion eventually associated with systemic chemotherapy if patient's general condition allows.

In a early-disseminated tumor cells profile, metastatic cells can accumulate alterations at a distant site and have a different profil from the original tumor cells. Metastatic cells can also accumulate alterations in the course if systemic treatments. Consequently, they may respond differently to drugs.

Recently, EGFR mutations and ALK status discordance between primary tumors and pleural metastases have been demonstrated in a significant portion of lung adenocarcinomas. These studies, realized on malignant pleural effusion isolated cells, enabled us to hypothesize a possible intratumoral heterogeneity within pleural metastases, but no study has been carried out on pleural tissue.

Our aim is to create a biocollection with tissues from pleural carcinomatosis in order to subsequently allow multiomics and bioinformatics analyzes and to characterize a possible intratumoral heterogeneity in pleural metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Malignant pleural effusion with or without prior histological or cytological diagnosis
* Patient eligible for a pleural biopsy for diagnostic purposes and validated in a multidisciplinary consultation meeting
* Having given their free and informed writing consent
* Affiliated to a social security system or assimilated

Exclusion Criteria:

* Malignant pleural mesothelioma
* Contraindication to general anesthesia
* Pregnant or breastfeeding woman, or is of child bearing potential and who did not agree to use highly effective methods of birth control throughout the study.
* Patient participating in a interventional study likely to interfere with this study
* Patient benefiting from a legal protection measure (guardianship or curatorship)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adult patients with pleural metastasis eligible for a surgical exploration of the pleura
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Blood samples are collected and a piece of biopsy will be used for the constitution of a specific collection in the CRB (Centre de ressource biologique) | At Day 1: day of surgery
  Blood samples are collected and a piece of biopsy will be used for the constitution of a specific collection in the CRB (Centre de ressource biologique)

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Drevet, MD, Principal Investigator — Department of Thoracic Surgery - Louis Pradel Hospital
Locations (1):
- Louis Pradel Hospital, Bron, France